CLINICAL TRIAL: NCT04217720
Title: An Open-Label, Multi-Center Phase 2 Clinical Trial Evaluating SNS-301 in Patients With ASPH+ High Risk Myelodysplastic Syndrome and Chronic Myelomonocytic Leukemia
Brief Title: SNS-301 Monotherapy in High Risk MDS and CMML
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Sensei Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNS-301-2-1
Record Dates: First submitted 2019-10-31; First posted 2020-01-03 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia (CMML)
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SNS-301 (Experimental): SNS-301
  Interventions: Drug: SNS-301

INTERVENTIONS:
Drug: SNS-301 — SNS-301 (1x 1011 dose/1ml) ID injection every 3 weeks for 4 doses then every 6 weeks for 6 additional doses, and thereafter every 12 weeks up to 24 months.

SUMMARY:
To evaluate safety, immunogenicity and anti-tumor responses of intradermally delivered SNS-301 in patients with ASPH+ high risk MDS and CMML.

DETAILED DESCRIPTION:
This phase 2, open-label, multi-center trial to evaluate the safety, immunogenicity and preliminary clinical efficacy of intradermally-delivered SNS-301 delivered using the 3M® hollow microstructured transdermal system (hMTS) device in patients with ASPH+ high risk myelodysplastic syndrome (MDS) and chronic myelomonocytic leukemia (CMML). The trial population consists of high risk ≥ Intermediate Risk-3 (IR-3) MDS and CMML-2.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Be 18 years of age or older.
3. Confirmed diagnosis of MDS or CMML.
4. Assessment of high-risk-MDS/CMML status defined as follows:

   1. MDS: IPSS-R criteria for categorization ≥ Intermediate Risk-3
   2. CMML: WHO criteria for CMML-2 (peripheral blasts of 5% to 19%, and 10% to 19% bone marrow blasts and/or presence of Auer rods).
5. Be willing to provide a fresh bone marrow aspirate sample at pre-treatment and demonstrate ASPH expression by flow cytometry.
6. Patient who has relapsed or is refractory / intolerant of hypomethylating agents (HMAs) or not responding to 4 treatment cycles of decitabine or 6 treatment cycles of azacytidine or progressing at any point after initiation of an HMA.
7. Patient refuses or is not considered a candidate for intensive induction chemotherapy using consensus criteria for defining such patients.
8. Patients with CMML must have been treated with at least 1 prior therapy (hydroxyurea or an HMA).
9. Eastern Cooperative Oncology Group (ECOG) Performance Scale 0-1.
10. Demonstrate adequate organ function: renal, hepatic, coagulation parameters.
11. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use two highly effective contraceptive methods during the treatment period and for at least 180 days after the last dose of study treatment. For male patients: Agree that during the period specified above, men will not father a child. Male patients must remain abstinent, must be surgically sterile during the treatment period and for at least 180 days after the last dose of study treatment.

Exclusion Criteria:

1. Any approved anti-cancer therapy including chemotherapy, targeted small molecule therapy or radiation therapy within 2 weeks prior to trial Day 0.
2. Participated on a clinical trial of an investigational agent and/or investigational device within 28 days prior to Day 0.
3. Malignancies other than indications open for enrollment within 3 years prior to Day 0.
4. Diagnosis of a core binding factor leukemia (t(8;21), t(16;16); or inv(16)) or diagnosis of acute promyelocytic leukemia (t(15;17)).
5. Active or history of autoimmune disease or immune deficiency.
6. History of HIV. HIV antibody testing recommended per investigator's clinical suspicion.
7. Active hepatitis B (hepatitis B surface antigen reactive) or active hepatitis C (HCV qualitative RNA detected); testing recommended per investigator's clinical suspicion.
8. Severe infections within 4 weeks prior to enrollment.
9. Received therapeutic oral or IV antibiotics within 2 weeks prior to Day 0.
10. History or current evidence of any condition, therapy or laboratory abnormality that in the opinion of the treating investigator might confound the results of the trial.
11. Known previous or ongoing, active psychiatric or substance abuse disorders that would interfere with the requirements of the trial.
12. Treatment with systemic immunomodulating agents (including but not limited to IFNs, IL-2) within 6 weeks or five half-lives of the drug, whichever is shorter, prior to first dose.
13. Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events of SNS-301 | 12 weeks
  Number of adverse events including adverse events of special interest as assessed by CTCAE v5.0
Objective response rate by International Working Group (IWG) 2006 criteria | 12 weeks
  Best objective response during the study
Minimal residual disease by IWG 2006 criteria | 12 weeks
  Minimal residual disease by peripheral and bone marrow blast count during the study
Duration of Response by IWG 2006 criteria | 12 weeks
  Duration of response calculated from date of first response to date of progression
Disease control rate (DCR) by IWG 2006 criteria | 12 weeks
  Disease control rate calculated as the proportion of patients with stable disease or better
Progression Free Survival (PFS) as assessed by IWG 2006 criteria | 12 weeks
  Progression free survival calculated from the date of start of treatment to date of progression
Overall Survival | 36 months
  Overall survival calculated from date of treatment to date of death

SECONDARY OUTCOMES:
Measurement of ASPH specific responses | up to 12 weeks
  Evaluate blood and tissue ASPH-specific responses at pretreatment, changes during treatment and at progression or end of study in all study participants where sample is available for analysis
Measurement of T cell immune response | up 12 weeks
  Characterize blood and bone marrow T cell types and numbers at pretreatment, changes during treatment and at progression or end of study in all study participants where sample is available for analysis
Measurement B cell immune responses | up to 12 weeks
  Characterize blood and bone marrow B cell numbers at pretreatment, changes during treatment and at progression or end of study in all study participants where sample is available for analyses
Evaluation of immune gene transcript profiles | up to12 weeks
  Determine changes in commercially available gene signature panels in blood and bone marrow pretreatment, during treatment and at progression in all study participants where sample is available for analysis
Measurement of pro-inflammatory and/or immunosuppressive molecules | up to 12 weeks
  The immunological response of pro-inflammatory/immunosuppressive molecules will be observed before, during and after treatment using commercially available assays. Analyses will be performed both on blood and bone marrow samples in all study participants where sample is available for analysis
Measurement of oncoprotein expression | up to 12 weeks
  Changes in oncoprotein levels will be evaluated before, during and after treatment using methods such as flow cytometry. Analyses will be performed both on blood and bone marrow samples in all study participants where sample is available for analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ildiko Csiki, MD, PhD, Study Director — Sensei Biotherapeutics

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results reported in the article, after deidentification (text, tables, figures and appendices) will be shared to researchers who have provide a methodologically sound proposal and sign a data access agreement.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Access will be considered to researchers who provide a methodologically sound proposal. Analysis must achieve the aims outlined in the approved proposal Proposals should be directed to info@senseibio.com. To gain access, data requestors will need to sign a data access agreement. Data are available for 36 months following article publication.